CLINICAL TRIAL: NCT04633889
Title: Deferoxamine for the Prevention of Cardiac Surgery-Associated Acute Kidney Injury
Acronym: DEFEAT-AKI
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David Leaf, Associate Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020P003605; R01DK125786 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-11-18 (Actual); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Deferoxamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Deferoxamine (Experimental): Deferoxamine 30mg/kg (max dose, 6g) intravenous infusion (diluted in 240mL normal saline) administered over 12 hours
  Interventions: Drug: Deferoxamine
- Placebo (Placebo Comparator): Normal saline (240mL) intravenous infusion over 12 hours
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Deferoxamine — Deferoxamine 30mg/kg (max dose, 6g) intravenous infusion (diluted in 240mL normal saline) administered over 12 hours
  Arms: Deferoxamine
Drug: Normal saline — Normal saline (240mL) intravenous infusion over 12 hours
  Arms: Placebo

SUMMARY:
Multiple lines of evidence support a central role of iron in causing acute kidney injury (AKI), including the finding that prophylactic administration of iron chelators attenuates AKI in animal models. Patients undergoing cardiac surgery may be particularly susceptible to iron-mediated kidney injury due to the profound hemolysis that often occurs from cardiopulmonary bypass. The investigators will test in a phase 2, randomized, double-blind, placebo-controlled trial whether prophylactic administration of deferoxamine decreases the incidence of AKI following cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Undergoing coronary artery bypass graft and/or valve surgery with cardiopulmonary bypass
3. AKI risk score ≥6 at the time of screening
4. Written informed consent from the patient or surrogate

Exclusion Criteria:

1. AKI, defined as any of the following:

   * Increase in serum creatinine ≥0.3 mg/dl in 48h
   * Increase in serum creatinine ≥50% in 7d (if no value available in last 7d, use most recent value in last 3 months)
   * Urine output ≤0.5 ml/kg/h x 6 consecutive hours (only assessed in patients with hourly monitoring via Foley catheter)
   * Receipt of renal replacement therapy (RRT) within 7d
2. Advanced chronic kidney disease (eGFR <15 ml/min/1.73m2 or end-stage kidney disease receiving RRT)
3. Hemoglobin <8 g/dL (closest value in the prior 3 months)
4. Fever (temperature ≥38⁰C) in the last 48h
5. Suspected or confirmed bacteremia, endocarditis, or pyelonephritis
6. Pneumonia, aspiration, or bilateral pulmonary infiltrates from an infectious etiology reported on chest x-ray or CT scan in the last 7d
7. Positive COVID-19 test within previous 10d
8. Chronic iron overload (including conditions such as hemochromatosis and beta thalassemia major) or previous iron chelation therapy (including prior participation in DEFEAT-AKI)
9. Known hypersensitivity to deferoxamine
10. Taking prochlorperazine
11. Severe hearing loss
12. Pregnant or breastfeeding
13. Prisoner
14. Concurrent participation in another interventional research study in which the intervention has potential interaction with deferoxamine
15. Surgery to be performed under conditions of circulatory arrest
16. Receiving extracorporeal membrane oxygenation
17. Durable ventricular assist device (VAD) prior to surgery (does not include Impella device or intra-aortic balloon pump)
18. Any condition which, in the judgement of the investigator, might increase the risk to the patient
19. Conflict with other research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2026-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David E. Leaf, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma S, Leaf DE. Iron Chelation as a Potential Therapeutic Strategy for AKI Prevention. J Am Soc Nephrol. 2019 Nov;30(11):2060-2071. doi: 10.1681/ASN.2019060595. Epub 2019 Sep 25. PMID 31554656
- [Derived] Scurt FG, Bose K, Mertens PR, Chatzikyrkou C, Herzog C. Cardiac Surgery-Associated Acute Kidney Injury. Kidney360. 2024 Jun 1;5(6):909-926. doi: 10.34067/KID.0000000000000466. Epub 2024 May 1. PMID 38689404

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The discrepancy between the number of patients enrolled (n=320) versus the number randomized, dosed, and included in the final analysis (n=301) was due to some patients being withdrawn from the study after enrollment but prior to randomization.
Groups:
- Deferoxamine: Deferoxamine 30mg/kg IV infusion x 12 hours starting preoperatively; Maximum total dose, 6g
- Placebo: Saline IV infusion x 12 hours starting preoperatively
Period: Overall Study
Arm/Group | Deferoxamine | Placebo
Started | 151 | 150
Completed | 151 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Deferoxamine | Placebo | Total
Number analyzed (Participants) | 151 | 150 | 301
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [63 to 75] | 70 [62 to 76] | 70 [63 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 36 | 81
  Male | 106 | 114 | 220
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 134 | 139 | 273
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 17
  Not Hispanic or Latino | 143 | 140 | 283
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Acute Kidney Injury
Description: Composite outcome that includes any of the following:
  1. Urine output <0.5 ml/kg/h for ≥6 consecutive hours within the first 48h or until the Foley catheter is removed, whichever occurs first
  2. Increase in serum creatinine ≥0.3 mg/dl within the first 48h
  3. Increase in serum creatinine ≥50% within 7 days
  4. Receipt of renal replacement therapy within 7 days
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Participants | 99 | 108
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.23, Chi-squared

2. Secondary Outcome: Renal Tubular Injury
Description: Urine levels of KIM-1
Time Frame: 3 days
Reporting Status: Not Posted, anticipated posting 2026-03

3. Secondary Outcome: Number of Participants With Major Adverse Kidney Events
Description: Defined as an increase in serum creatinine ≥100%, receipt of renal replacement therapy, or death within 7 days
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Participants | 14 | 13

4. Secondary Outcome: Number of Participants With Postoperative Myocardial Injury
Description: Defined as postoperative hs-cTnI concentration ≥ the 90th percentile of the cohort on either postoperative day 1 or 2.
Time Frame: 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Participants | 15 | 15

5. Secondary Outcome: Number of Participants With Atrial Fibrillation or Atrial Flutter
Description: Defined as new onset postoperative atrial fibrillation or atrial flutter (patients with atrial fibrillation or atrial flutter at baseline will be excluded)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 102 | 90
Participants | 33 | 32

6. Secondary Outcome: Number of Participants With Prolonged Mechanical Ventilation
Description: Defined as a requirement for mechanical ventilation >24h postoperatively
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Participants | 31 | 27

7. Secondary Outcome: Time to Liberation From Vasoactive Medications
Description: Number of hours from time of incision to liberation from all IV vasoactive medications
Time Frame: 7 days
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Hours | 29 [20 to 59] | 30 [15 to 50]

8. Secondary Outcome: Number of Participants With Sepsis
Description: Defined as a life-threatening organ dysfunction caused by a dysregulated host response to infection. Organ dysfunction is defined as an acute increase in the total SOFA score ≥2 points consequent to the infection.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Participants | 6 | 2

9. Secondary Outcome: Ventilator-free Days
Description: 28 minus the number of days ventilated. Patients who die within 28 days will be assigned 0 ventilator-free days.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Days | 27 [27 to 28] | 28 [27 to 28]

10. Secondary Outcome: ICU-free Days
Description: 28 minus the number of days in the ICU. Patients who die within 28 days will be assigned 0 ICU-free days.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Days | 25 [23 to 26] | 25 [23 to 26]

11. Secondary Outcome: Hospital-free Days
Description: 28 minus the number of days hospitalized. Patients who die within 28 days will be assigned 0 hospital-free days.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Deferoxamine | Placebo
Number analyzed (Participants) | 151 | 150
Days | 20 [16 to 22] | 20 [14 to 22]

ADVERSE EVENTS:
Time Frame: All-cause mortality was measured from initiation of the study drug until discharge from the index hospital admission during which the study drug was administered, up to 1 year; Vasoactive-Inotropic Score (VIS) was measured for 24-hours following study drug initiation; anaphylaxis was measured throughout the 12 hour study drug administration period; Infection/Sepsis and ARDS were measured for 7 days following the study drug administration.
Description: We limited the scope of our adverse events (AEs) monitoring and reporting to a prespecified list of AEs of special interest (AESI)-anaphylaxis, infection/sepsis, VIS ≥ 30, and ARDS-since the patient population was undergoing high risk surgery and it was expected that they would have a number of unrelated adverse health events during the course of their hospital stay.
Arm/Group | Deferoxamine | Placebo
All-Cause Mortality (participants affected / at risk) | 6/151 | 6/150
Serious Adverse Events (participants affected / at risk) | 23/151 | 25/150
Other Adverse Events (participants affected / at risk) | 0/151 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Deferoxamine (N=151) | Placebo (N=150)
Anaphylaxis (Immune system disorders) | 0 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Infection/Sepsis (Infections and infestations) | 12 | 8
Vasoactive-Inotropic Score ≥30 (Cardiac disorders) | 17 | 21 — The Vasoactive-Inotropic Score (VIS) is a linear composite of vasoactive and inotropic infusion rates. Higher scores indicate greater hemodynamic support, with 0 as the minimum and values ≥30 indicating profound cardiovascular failure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT04633889/Prot_SAP_000.pdf